CLINICAL TRIAL: NCT02909933
Title: Low Dose Liraglutide and Metformin vs. High Dose Liraglutide Alone in Treatment of Obesity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Andrej Janez, MD PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COMBO - LIRA 3
Record Dates: First submitted 2016-09-13; First posted 2016-09-21 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2015-06

CONDITIONS: Polycystic Ovary Syndrome; Obesity
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity | interventions — Liraglutide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- liraglutide (Experimental): liraglutide 3 mg QD for 12 weeks
  Interventions: Drug: liraglutide
- metformin and liraglutide (Experimental): metformin 1000 mg BID and liraglutide 1.2 mg QD for 12 weeks
  Interventions: Drug: metformin and liraglutide

INTERVENTIONS:
Drug: liraglutide
  Other Names: Victoza
  Arms: liraglutide
Drug: metformin and liraglutide
  Other Names: Glucophage and Victoza
  Arms: metformin and liraglutide

SUMMARY:
Weight reduction is the most important treatment target when polycystic ovary syndrome (PCOS) is linked to obesity. Liraglutide (LIRA) in dose of 3 mg was recently approved as an anti-obesity drug. Metformin could enhance weight lowering potential of liraglutide.

We investigates short term interventions with low dose liraglutide in combination with metformin and high dose liraglutide alone influence on significant weight reduction in obese women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old to menopause
* polycystic ovary syndrome (NICHD criteria)
* BMI of 30 kg/m² or higher

Exclusion Criteria:

* type 1 or type 2 diabetes mellitus
* history of carcinoma
* Cushing's syndrome or congenital (non-classic) adrenal hyperplasia
* personal or family history of MEN 2
* significant cardiovascular, kidney or hepatic disease
* the use of medications known or suspected to affect reproductive or metabolic functions
* the use of statins, within 90 days prior to study entry

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The main outcome was change in body weight. | Patient's body weight was measured at the base point and after 12 weeks of clinical trial.

SECONDARY OUTCOMES:
The secondary outcome was change in body mass index (BMI) | Patient's body weight were measured at the base point and after 12 weeks of clinical trial. Patient's height was measured at the base point.

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Janez, MD PhD, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Medical Center Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jensterle M, Kravos NA, Goricar K, Janez A. Short-term effectiveness of low dose liraglutide in combination with metformin versus high dose liraglutide alone in treatment of obese PCOS: randomized trial. BMC Endocr Disord. 2017 Jan 31;17(1):5. doi: 10.1186/s12902-017-0155-9. PMID 28143456